CLINICAL TRIAL: NCT01254162
Title: A 4-Week, Randomized, Double-Blind, Placebo-Controlled Proof-of-Concept Study to Evaluate the Potential of Topically Applied 0.75% (w/w) MTC896 Gel to Reduce Sebum Production on the Forehead of Healthy Male Volunteers
Brief Title: Proof of Concept Study of MTC896 Gel to Reduce Sebum Production on the Forehead of Healthy Male Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mimetica Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCL10001
Record Dates: First submitted 2010-12-02; First posted 2010-12-06 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Oily Skin; Seborrhea
Keywords: Oily Skin; Sebum
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Placebo Gel (Experimental)
  Interventions: Drug: MTC896 Gel

INTERVENTIONS:
Drug: MTC896 Gel — 0.75% w/w gel applied daily for 28 days to the forehead

SUMMARY:
To determine the potential of topically applied 0.75% (w/w) MTC896 Gel to reduce sebum production on the forehead of healthy male volunteers.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled proof-of-concept study of the investigational product (0.75% (w/w) MTC896 Gel) compared to a placebo control. Subjects will be randomized to 1 of 2 treatment groups, 0.75% (w/w) MTC896 Gel or Placebo. Approximately 134 subjects will be enrolled to yield 60 completed subjects in each group. One group will receive once daily topical applications of 0.75% (w/w) MTC896 Gel to the forehead for 28 consecutive days, and the other will receive placebo under the identical regimen. Enrollment will be staggered to allow monitoring of safety and tolerability. A lead cohort will include approximately 20 subjects (10 in the MTC896 Group and 10 in the Placebo Group). Application on additional subjects will not be initiated until the lead cohort has completed the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Are healthy males;
* 2. Are between 18 and 65 years of age;
* 3. Have self-perceived oily skin confirmed by a clinical assessment;
* 4. Have an average Sebumeter® reading of ≥ 220 µg/cm2 on the forehead;
* 5. Have a negative urine drug screening test result;
* 6. Have a negative HIV and hepatitis screening test result;
* 7. Agree to use adequate contraceptive precautions (ie, use of condoms) during the conduct of the study;
* 8. Have a body mass index (BMI) of 19 to 34 kg/m2;
* 9. Are free of any systemic or dermatologic disorder, which, in the opinion of the investigator, will interfere with the study results or increase the risk of adverse events;
* 10. Are willing to abstain from using any facial treatment products or personal care products (moisturizer, sunscreen, hair spray, etc) on the forehead during the study;
* 11. Are willing to avoid sun exposure and to protect the forehead with a hat/visor;
* 12. Are fluent in the English language;
* 13. Complete a standard Medical Screening form as well as a Medical Personal History form; and
* 14. Read, understand, and provide a signed informed consent.

Exclusion Criteria:

* 1. Have any visible skin disease at the application site which, in the opinion of the investigator, will interfere with the study evaluations;
* 2. Have a history of photosensitive reactions or a history of cutaneous or systemic lupus or other disorders frequently associated with photosensitivity;
* 3. Are not willing to refrain from using systemic/topical analgesics such as aspirin (81 mg daily aspirin will be allowed at the discretion of the PI), Aleve, Motrin, Advil, or Nuprin for 24 hours prior to and during the study (use of acetaminophen will be permitted);
* 4. Are using systemic/topical corticosteroids in the test area for 3 weeks prior to and during the study, or systemic/ antihistamines for 24 hours prior to and during the study;
* 5. Are using topical retinoids, products containing benzoyl peroxide, salicylic acid, or alpha-hydroxy acids for 2 weeks prior to and during the study; or systemic retinoids within 3 months prior;
* 6. Are using any medication which, in the opinion of the investigator, will interfere with the study evaluations;
* 7. Have seborrheic dermatitis and/or active atopic dermatitis/eczema in or around the test sites;
* 8. Have a known allergy and/or hypersensitivity to constituents present in the study products;
* 9. Have damaged skin in or around the test sites, including sunburn, excessively deep tans, uneven skin tones, tattoos, scars, excessive hair, numerous freckles, or other disfigurations of the test site;
* 10. Have received treatment for any type of internal cancer within 5 years prior to study enrollment;
* 11. Have a history of, or are currently being treated for skin cancer;
* 12. Are currently participating in any clinical testing; and/or
* 13. Have received any investigational treatment(s) within 4 weeks prior to study enrollment.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
A 20% reduction in sebum production as measured by the Sebumeter | 28 days

SECONDARY OUTCOMES:
Assess the safety and tolerability of the product when applied daily to the forehead for 28 days | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Dosik, MD, Principal Investigator — TKL Research, Inc.
Locations (1):
- TKL Research, Inc, Paramus, New Jersey, United States